CLINICAL TRIAL: NCT05559346
Title: Investigation of the Effects of Diaphragm Exercises in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Berna Karamancıoğlu, Research Assistant, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP1
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Palsy Spastic Diplegia
Keywords: cerebral palsy; respiratory strength; pulmonary functions; sitting ability
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research Group (Experimental): Diplegic Cerebral Palsy
  Interventions: Other: Diaphragmatic exercises
- Control Group (Active Comparator): Diplegic Cerebral Palsy
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Other: Diaphragmatic exercises — Diaphragm exercises will be applied to the research group in addition to conventional rehabilitation.The content of the individualized conventional rehabilitation program consists of passive stretching exercises, strengthening exercises to antagonists of spastic muscles and exercises aimed at improving weight transfer, balance and correction reactions, and postural control. In addition to conventional rehabilitation, manual diaphragmatic relaxation exercises and diaphragmatic breathing exercises will be applied to the children in the research group two days a week.
  Arms: Research Group
Other: conventional physiotherapy — The control group will only be taken to the conventional rehabilitation program. e content of the individualized conventional rehabilitation program consists of passive stretching exercises, strengthening exercises to antagonists of spastic muscles and exercises aimed at improving weight transfer, balance and correction reactions, and postural control.
  Arms: Control Group

SUMMARY:
The aim of this study is to examine the effects of diaphragmatic myofascial relaxation exercise and diaphragmatic breathing exercises added to the conventional physiotherapy and rehabilitation program in children with diplegic cerebral palsy (CP), primarily on MIP, MEP, and secondarily on thoracic cage mobility, pulmonary functions and sitting ability.

DETAILED DESCRIPTION:
This research is a randomized controlled trial. Volunteers diagnosed with cerebral palsy who applied to Marmara University Pendik Training and Research Hospital will participate in the research. A voluntary consent form will be obtained from the participants at the beginning of the study. Demographic and clinical information form will be filled for each patient at the beginning of the study before clinical evaluations. Demographic and clinical information form; Age, gender, height, weight, body mass index (BMI), how many weeks were born, birth weight, drug use, disease history, number of siblings, neonatal intensive care hospitalization history, education level of parents will be questioned. The Gross Motor Functional Classification System (KMFSS) will be used to determine the functionality levels of the volunteers who will participate in the study. The following tests will be applied to all of the volunteers who will participate in our study before and after the intervention:

Respiratory Muscle Strength Measurement Thoracic Cage Mobility Assessment Pulmonary Function Tests Gross Motor Functional Measurement (part B) Children meeting the inclusion criteria will be randomly assigned to two groups. The control and research groups will receive an individualized conventional rehabilitation program for 45 minutes, 2 days a week for 8 weeks. In addition to conventional rehabilitation, manual diaphragmatic relaxation exercises and diaphragmatic breathing exercises will be applied to the children in the research group two days a week.

After 8 weeks of intervention and control group applications, the evaluations made at the beginning of the intervention will be repeated. The evaluations of the two groups will be compared statistically and the results will be interpreted.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with spastic diplegic cerebral palsy
* Being between the ages of 5-15
* Gross Motor Functional Classification System 1,2 or 3
* To be at a cognitive level to be able to understand and apply the instructions in the tests (SFT, MIP, MEP) to be applied

Exclusion Criteria:

* Having had a surgical operation in the last 6 months
* Presence of scoliosis detected above 30 degrees
* Having a planned surgery within 3 months from the start of the study
* Have a chronic lung disease

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Respiratory Muscle Strength Measurement (Maximum inspiratory pressure) | 8 weeks
  It will be used as the primary outcome measure in the study. In our study, respiratory muscle strength will be measured with a portable intraoral pressure measuring device (MicroRPM) Maximum static inspiratory pressure (MIP) will be measured at residual volume after maximum expiration. Measurements will be made twice in a sitting position with verbal encouragement and using a nose clip. The highest value obtained, with no more than 10% or 10cmH2O difference between the two measured values, will be used for analysis
Respiratory Muscle Strength Measurement (Maximum Expiratory Pressure) | 8 weeks
  It will be used as the primary outcome measure in the study. In our study, respiratory muscle strength will be measured with a portable intraoral pressure measuring device (MicroRPM) Maximum static expiratory pressure (MEP) will be measured at maximum post-inspiratory total lung capacity.
  Measurements will be made twice in a sitting position with verbal encouragement and using a nose clip. The highest value obtained, with no more than 10% or 10 cmH2O difference between the two measured values, will be used for analysis
Thoracic Cage Mobility Assessment | 8 weeks
  Chest circumference measurements will be used to determine respiratory type. Measurements will be recorded in centimeters, using a tape measure, in an upright sitting position, from the axillary, epigastric and subcostal regions, the difference between neutral, deep inspiration and deep expiration

SECONDARY OUTCOMES:
Pulmonary Function Tests (PFT) | 8 weeks
  Pulmonary function tests will be performed with a spirometer device in the evaluation of pulmonary capacity. Pulmonary function tests are maneuvers applied to measure lung functions using standard devices. In this thesis, forced vital capacity (FVC), forced vital volume in one second (FEV1), FEV1/FVC and peak expiratory flow (PEF) values will be examined with pulmonary function tests.
Gross Motor Functional Measurement (Part B) | 8 weeks
  Sitting skill will be evaluated with the sub-section B of the Gross Motor Function Measure (GMFM) test. Sitting, which is part B, consists of 20 items. The gross motor functions in these items are evaluated according to the degree of achievement of the function. Scoring is done on a Likert scale between 0 and 3 points. A score of 0 indicates that the activity could not be started at all, and 3 indicates that 90-100% of it can be done.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Kenıs Coskun, PhD, Study Director — Marmara University
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No